CLINICAL TRIAL: NCT06891781
Title: A Prospective, Multi-center, Randomized, Double-blind, Cross Over, Clinical Trial to Compare the Safety and Effectiveness of Adaptive Versus Conventional Stimulation in Levodopa- Responsive Parkinson's Disease Treated with Bilateral Deep Brain Stimulation of the Subthalamic Nucleus
Brief Title: Investigating Adaptive Deep Brain Stimulation in Parkinson's Disease Management
Acronym: ADVENT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Newronika (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NWK_Pivotal_aDBS-PV01
Record Dates: First submitted 2025-03-11; First posted 2025-03-24 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Parkinson Disease, Idiopathic
Keywords: Deep Brain Stimulation; Parkinson Disease; adaptive Deep Brain Stimulation; aDBS; conventional Deep Brain Stimulation; cDBS
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Intervention Model Description: It is a prospective, multi-center, randomized, double-blind, cross over clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- aDBS (Experimental): adaptive DBS (closed-loop DBS)
  Interventions: Device: Deep Brain Stimulation
- cDBS (Active Comparator): conventional DBS
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation — AlphaDBS System

SUMMARY:
The goal of this prospective, multi-center, randomized, double-blind, crossover clinical trial is to evaluate the effectiveness and safety of adaptive DBS (aDBS) and conventional DBS (cDBS) delivered through the AlphaDBS system, in levodopa-responsive Parkinson's disease subjects. Data from previous studies conducted in Europe indicate that the use of the AlphaDBS system is safe and effective in both aDBS and cDBS modes. However, such studies suggest that aDBS may lead to more ON-time without troublesome dyskinesias in some patients. The study is designed to first demonstrate safety of effectiveness of cDBS, then to directly compare effectiveness of aDBS relative to cDBS. Subjects enrolled in the study will undergo multiple visits to assess the improvement of PD symptoms and will be randomized to Mode 1 for three months, followed by Mode 2. At the end of Mode 2, subjects will select their preferred mode, which will be maintained for 3 additional months. Subjects will complete patient diaries at different time points to evaluate their symptoms throughout the day.

ELIGIBILITY:
INCLUSION CRITERIA

A subject who meet all of the following criteria may be given consideration for inclusion in this clinical trial:

* Is willing and capable of signing informed consent
* Is ≥18 years old
* Has been diagnosed with levodopa-responsive idiopathic Parkinson's disease
* Has a Hoehn and Yahr (H&Y) scale stage of II or III when OFF medication at screening
* Exhibits motor fluctuations and PD-related symptoms that are not adequately controlled with medication, including motor complications of recent onset (>4 months duration)
* Has been referred for bilateral STN DBS in accordance with local practice
* Must be a good surgical candidate for placement of a deep brain stimulator as judged by the DBS surgical team
* Montreal Cognitive Assessment score of ≥ 26 at the screening visit (when in "medON" state)
* UPDRS-III improvement by ≥30% with the levodopa challenge test as measured at approximately 90 minutes following administration of the challenge dose
* Successfully completed a 1-day test diary reaching a sufficient level of agreement (>75%) with study personnel responses and is willing and capable of completing a 5-day diary at each of the time points required per the protocol
* If female, the subject is not currently pregnant (as determined by negative serum pregnancy test), breastfeeding, or is post-menopausal, surgically sterile or willing to use birth control for the duration of the study - acceptable forms of birth control are: hormone therapies (oral, injected, transdermal or implanted), IUD or other barrier methods (e.g., condom, diaphragm, cervical cap, spermicide/gel) or partner is surgically sterile
* Is willing to maintain a constant anti-PD medication treatment (best medical management) for at least one month prior to DBS implantation
* Is willing and able to attend all study-required visits, complete the study procedures and attend appropriate follow-up visits

EXCLUSION CRITERIA

* Has contraindications for DBS surgery, including any intracranial abnormality (e.g., generalized atrophy, vascular malformation, hydrocephalus, hematoma, cavernous or venous angioma, tumor or metastases, midline shift, etc.) or metallic implant (e.g., aneurysm clip, cochlear implant, etc.) or other clinically significant space-occupying lesion which in the opinion of the surgeon would impact the ability to target and place the leads or IPG
* Is unable or unwilling to maintain a stable dose of levodopa anti-Parkinson's disease medication for 30 days prior to DBS surgery
* Has any current major psychiatric disorder(s), such as Major Depressive Disorder, Bipolar I or II disorder, Schizophrenia, Schizoaffective Disorder, Delusional Disorder, Brief Psychotic Disorder, Obsessive-Compulsive Disorder, or any other current psychiatric condition that in the opinion of the investigator would confound the assessment of study endpoints, prevent proper data collection and/or compromise the subject's ability to participate, based on the psychiatric/psychological assessment at screening. It refers also to moderate or severe alcohol and/or substance use disorder based on the psychiatric/psychological assessment at screening. (It is permitted if a subject has a diagnosis of Major Depressive Disorder with symptoms that currently are well-controlled and managed by a stable regimen of antidepressants for a minimum of 4 weeks prior to the screening visit).
* A history of suicide attempt within 3 years of the screening visit or current active suicidal ideation as determined by a psychiatric/ psychological evaluation
* Any medical condition, such as cognitive impairment, dementia, seizures, congestive heart failure, unstable angina, uncontrolled diabetes, renal failure requiring dialysis, or any other severe medical condition that could interfere with study procedures, confound the assessment of study endpoints, prevent proper data collection, or that, in the opinion of the investigator, would compromise the subject's ability to participate
* Confirmation of diagnosis of a terminal illness associated with survival <12 months
* Needs repeated MRI scans
* Requires diathermy, transcranial magnetic stimulation (TMS), or electroconvulsive therapy (ECT)
* Has an electrical or electromagnetic implant (e.g., cochlear prosthesis, pacemaker, neurostimulator, etc.) or plans to obtain, an active implanted medical device (AIMD) and/or an implanted medication pump (e.g., DUOPA™ infusion pump) and/or is treated with a portable infusion pump for any indication
* Is on anticoagulant therapy which cannot be paused for >5 days before surgery
* A history of cranial surgery including ablation procedure or any other previous neurosurgical procedure for the treatment of PD symptoms on either side of the brain
* Is currently participating in another clinical study (excluding any sub-study of the present trial).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Improvement in Good On Time (GOT) | After 3 months of follow up in cDBS as compared with pre-op baseline
  Mean improvement in GOT with conventional DBS (cDBS), when compared with pre-operative baseline

SECONDARY OUTCOMES:
GOT difference between aDBS and cDBS | After 3 months of follow up in each mode
  The mean difference in GOT (aDBS - cDBS) at the end of the second crossover period
UPDRS III score difference between aDBS and cDBS | After 3 months of follow up in each mode
  The mean difference in UPDRS III scores (aDBS - cDBS) at the end of the second crossover period
PDQ-39 score difference between aDBS and cDBS | After 3 months of follow up in each mode
  The mean difference in PDQ-39 score (aDBS - cDBS) at the end of the second crossover period
Subject Preference for aDBS vs. cDBS | After 3 months of follow up in each mode
  The proportion of subjects that prefer adaptive mode over conventional mode, according to subject preference selection
Comparison of Subject Preference for aDBS vs. cDBS based on PGI-I Ratings | After 3 months of follow up in cDBS as compared with pre-op baseline
  Proportion of subjects rating aDBS higher than cDBS when reporting on the PGI-I

OTHER OUTCOMES:
Assessment of time to symptom relief in aDBS vs cDBS | After 3 months of follow up in each mode
  aDBS reduces time to symptom relief faster than cDBS
Users feedback on the AlphaDBS System | After 3 months of follow up in each mode
  Users feedback on the AlphaDBS System evaluated through questionnaires in which the patients and the physicians are required to score their satisfaction in relation to the easiness of use of selected device features (from 1, minimum score to 5, maximum score).
AlphaDBSipg functionality | After 3 months of follow up in each mode
  * Local Field Potential (LFP) signals
  * Recharging (time, frequency, and number of cycles)
Resource utilization | From implant to the end of the study
  * The PDQ-39
  * Number and nature of participant communications by phone or messaging to the treating neurologist for problems related to PD or trial participation
  * Number and duration of healthcare visits (outsubject clinic, emergency unit, or hospital admission) for issues related to PD or clinical trial participation
Neurophysiologic signal quality and stability | From implant to the end of the study
  * Number of hemispheres with detectable beta power
  * Cardiac and other artifact occurrence
Safety Objectives | From screening till the end of the study
  * Incidence of adverse events from implantation through each crossover period.
  * All adverse events occurring during the entire duration of the study will be collected and reported.
  * Acute safety will evaluate all procedure-related adverse events occurring through the first 30 days post-implant.
  * Long-term safety of the implant will evaluate all procedure- and device-related adverse events occurring between 30 days and the conclusion of Mode 2 post implant.
  * Therapy safety will evaluate all therapy-related adverse
  * Events occurring between 30 days and the conclusion of Mode 2 post implant.
Fluctuations in disease symptoms | After 3 month of follow up in each mode
  Number of ON/OFF transitions based on the 3-day diary
Concomitant use of anti-parkinsonian medications | After 3 month of follow up in each mode
  Number of levodopa dose equivalents
Mentation, behavior and mood | After 3 month of follow up in each mode
  Evaluation of mentation, behavior, and mood through UPDRS (Unified Parkinson's Disease Rating Scale) part I.
  Minimum value 0 (best) and maximum value 52 (worst).
Activities of daily life (ADLs) | After 3 month of follow up in each mode
  Evaluation of the activities of daily life (ADLs) including speech, swallowing, handwriting, dressing, hygiene, falling, salivating, turning in bed, walking, and cutting food through UPDRS (Unified Parkinson's Disease Rating Scale) part II. Minimum value 0 (best) and maximum value 52 (worst).
Complications of therapy | After 3 month of follow up in each mode
  Evalutation of complications of therapy through UPDRS (Unified Parkinson's Disease Rating Scale) part IV. Minimum value 0 (best) and maximum value 24 (worst).
Capabilities of people with impaired mobility | After 3 month of follow up in each mode
  Assessment of capabilities of people with impaired mobility through Schwab and England Scale (SE). Minimum value 0% (worst) and maximum value 100% (best).
Cognitive impairment | After 3 month of follow up in each mode
  Evaluation of cognitive impairment through Montreal Cognitive Assessment (MoCA). Maximum value 30 (normal ≥ 26)
Freezing of Gait (FOG) severity | After 3 month of follow up in each mode
  Assessment of FOG severity through Freezing of Gait Questionnaire (FOG-Q). Minimum value 0 (best) and maximum value 24 (worst)
Balance | After 3 month of follow up in each mode
  Assessment of balance through Mini Balance Evaluation Systems Test (MiniBEST) which consists of four tasks divided into four subcomponents: anticipatory postural adjustments, postural responses, sensory orientation and dynamic gait.
Movement of Hands and Arms | After 3 month of follow up in each mode
  Hand-Arm movement test in stimON/medOFF and stimON/medON condition is used to evaluate subjects capability to move hands and arms.
Mobility | After 3 month of follow up in each mode
  Subject's mobility evaluated through Timed Up and Go test in stimON/medOFF and stimON/medON condition
Quality of life assessment | After 3 month of follow up in each mode
  Subject's quality of life will be assessed through a self-assessment questionnaire (EQ-5D-5L).
Health related quality of life assessment | After 3 month of follow up in each mode
  Subject's health related quality of life will be assessed through the Short Form Health Surve (SF-36) questionnaire. Minimum value 0 (worst) and maximum value 100 (best)
Non-motor symptoms associated with Parkinson's disease | After 3 month of follow up in each mode
  Non-motor symptoms associated with Parkinson's disease will be evaluated through PD Non-motor symptom Self-Assessment questionnaire. Each symptom scored with respect to: severity (0=none;1=mild;2=moderate;3=severe) and frequency (1=rarely;2=often;3=frequent;4=very frequent). Yes/no answers are not included in final frequency x severity calculation.
Clinician Global Impression | After 3 month of follow up in each mode
  The Clinician Global Impression (CGI) scale is a standardized assessment scale for determining the effects of mental health treatment. The scale is divided into CGI- S to evaluate the severity of illness and CGI-I to evaluate the improvement. Minimum value 0 (best) and maximum value 7 (worst)